CLINICAL TRIAL: NCT02321735
Title: The Genomic, Epigenomic, and Psychosocial Characteristics of Long-Term Survivors of Ovarian Cancer - Recruitment
Brief Title: DOD Long-Term Survivors of Ovarian Cancer
Acronym: LTSOC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Michael J. Birrer,M.D.,Ph.D., Director, Gynecologic Medical Oncology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2014P000798; W81XWH-13-1-0413 (Other Grant/Funding Number: DOD)
Record Dates: First submitted 2014-12-17; First posted 2014-12-22 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Ovarian Cancer
Keywords: Long-Term Survivor; Genomic; Survivorship; Quality of Life
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Long-Term Ovarian Cancer survivors (Other): Genomic, immunologic and psychosocial characterization of Long-Term survivors of ovarian cancer. This will involve a Quality of Life Questionaire.
  Interventions: Behavioral: Quality of life questionaire

INTERVENTIONS:
Behavioral: Quality of life questionaire — Patients will participate in a QOL questionaire followed by a phone interview

SUMMARY:
: Stages III and IV serum ovarian cancer are the most lethal of all gynecologic cancers; however, some advanced-stage ovarian cancer patients are long-term survivors. These patients may provide the key to long-term survival and bring hope to all women with Stages III and IV ovarian cancer. There is no meaningful explanation of why some patients with ovarian cancer become long-term survivors and what their quality of life is long after their initial diagnosis. This research project will specifically determine molecular features within tumors along with genetic, quality of life, and lifestyle features that predict for long-term survival for patients with Stages III and IV ovarian cancer. It will bring together sophisticated molecular techniques, researchers with longstanding interest, a wide spectrum of consumer advocates (a number being long-term survivors), and quality of life experts to analyze the most carefully maintained patient database in the world-the Gynecologic Oncology Group database. We anticipate the results from this project will identify specific biochemical pathways and genetic features associated with long-term survival that can be used to improve the treatment, survival, and survivorship of patients with this disease. There is clearly something unique among patients who survive Stage III or IV ovarian cancer long term, and we believe that when we understand what this is, we can increase the number of long- and longer-term survivors.

DETAILED DESCRIPTION:
Background: Ovarian cancer (OC) remains a major health problem in the United Sates (US). In 2012, there will be an estimated 22,280 cases of epithelial OC (EOC) resulting in 15,500 deaths. While the median survival of OC patients has improved over the last two decades, the vast majority of patients suffer relapse and develop chemo-resistant disease. The overall survival of patients suffering from OC has not changed appreciably over the last three decades. Despite these dismal statistics, there is a minority of OC patients who are long-term (LT) survivors (>10 years). This includes a subset of advanced stage (~15%) and a higher proportion of early-stage disease (75%). Unfortunately, there is little genomic or biologic characterization of these tumors, or patient-reported outcomes that characterize LT survivors. The clinical importance of identifying subsets of patients who may or may not benefit from therapy, and understanding the biology of their tumors, is significant both from a patient survival and quality of life (QOL) standpoint. The characterization of LT survivors of advanced stage OC will potentially identify molecular and clinical pathways that can be targeted to help women who have shorter survivals. Further, careful characterization of these patients, including their initial and longitudinal health-related QOL reports, their response to treatments, and their tumors will provide significant measures of prognostic factors. Accurate identification of women with high-grade, early stage OC who will recur will allow for tailoring therapy to only those who will benefit. Thus, the systematic molecular and patient-reported outcomes evaluation of LT survivors of OC (both early and advanced stage) will yield data, which can significantly impact the management of OC patients.

Overall Aim: To characterize the genomic, biologic, and biobehavioral basis for LT survivors of EOC. We hypothesize that LT survivors of OC have distinct features that distinguish them from short-term (ST) survivors.

Specific Aims

1. To characterize the genomic, biologic, and immunologic features of tumors from LT versus ST survivors of advanced stage EOC. We propose to evaluate the genomic features (copy number variation, miRNA and methylation patterns) in LT (>7 years) versus ST survivors (<2 years). In addition, all cases will be evaluated for tumor infiltrating lymphocytes (TILs). Correlations between TILs and genomic parameters will be examined along with the identification of genomic/immune signatures that predict for LT survival. This aim leverages ongoing funded projects characterizing the transcriptome of advanced stage OC using GOG trials.
2. To validate a genomic signature that predicts for recurrence of early-stage, high-grade EOC. This aim will leverage an ongoing DOD grant (DOD#OC110628; Birrer, PI) generating a genomic signature (transcriptome) that distinguishes recurrent from non-recurrent early-stage, high-grade EOC.
3. To determine the extent to which health-related QOL measures, additional patient-reported outcomes (PROs), and key CTCAE criteria predict LT ovarian cancer survival.
4. To examine as an exploratory aim, the potential relationship between health-related QOL, PROs, and key CTCAE criteria with genomic features predicting disease recurrence.

Proposed Consortium: We propose utilizing the Gynecologic Oncology Group (GOG) infrastructure as the basis for the consortium, supplemented by the addition of research sites, administrative structure, advisory boards, and biostatistical support. We consider this to be a major advantage for this proposal in that the de novo creation of a consortium will not be necessary. GOG is the world's leading clinical trial organization focused on the prevention, diagnosis, and treatment of gynecologic cancers. GOG includes over 391 medical institutions participating in GOG clinical trials. As such, these institutions are familiar with all GOG procedures including the accurate collection of clinical and QOL data and the procuring and processing of tissue specimens. GOG institutions have extensive infrastructure in place to conduct large-scale clinical research and will serve as an established network of key sites for this project.

ELIGIBILITY:
Inclusion Criteria:

* stage III/IV high grade epithelial ovarian cancer diagnosed at least 10 years ago

Exclusion Criteria:

* early stage, low grade ovarian cancer diagnosed less than 10 years ago

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2014-09; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Quality of life questionnaire | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Birrer, MD PhD, Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital (The General Hospital Corp), Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
the study is still at a very early stage to understand how data will be shared